CLINICAL TRIAL: NCT04392635
Title: Pilot Study to Establish Safety and Ease of Use of a TauTona Pneumoperitoneum Assist Device (TPAD) for Laparoscopic Surgery
Brief Title: Device to Assist With Abdominal Access During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: TauTona Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-55013; NCT06361849 (obsolete NCT alias)
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TauTona Pneumoperitoneum Assist Device (TPAD) (Experimental): Participants will receive investigational TPAD device during laparoscopic surgery. The TPAD was used to aid Veress needle insertion in place of surgical tools such as clamps. The TPAD was applied to the patient prior to Veress needle entry and removed after insufflation was completed.
  Interventions: Device: TauTona Pneumoperitoneum Assist Device (TPAD)
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC included both direct (unassisted) entry and assisted entry using clamps, if needed, to aid in Veress needle insertion. Upon confirmation that the Veress needle was in the correct location (e.g. drop test), insufflation was initiated.
  Interventions: Procedure: Standard of Care (SOC)

INTERVENTIONS:
Device: TauTona Pneumoperitoneum Assist Device (TPAD) — The TPAD is an experimental device used to assist with placement of Veress needle during laparoscopic surgery.
  Arms: TauTona Pneumoperitoneum Assist Device (TPAD)
Procedure: Standard of Care (SOC) — Standard of Care was used for Veress needle insertion.
  Arms: Standard of Care (SOC)

SUMMARY:
The purpose of this study is to assess the safety and ease of use of a TauTona Pneumoperitoneum Assist Device (TPAD) to assist with obtaining peritoneal access with a Veress needle, and for placing a primary trocar, during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Scheduled for laparoscopic surgery
* Able to understand and willing to sign a written informed consent form

Exclusion Criteria:

* Age < 18
* Any situation where blind, peri-umbilical passage of a Veress needle is contraindicated.
* Any situation where patients have suspected or confirmed intra-abdominal adhesions involving the peri-umbilical abdominal wall.
* Any situation where patients have a suspected or confirmed umbilical hernia or peri-umbilical ventral hernia.
* Any situation where there is not intact, uncompromised skin of the peri-umbilical region where the device is to be placed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Korndorffer Jr, MD MHPE FACS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): Participants receive SOC including direct (unassisted) entry and/or assisted entry using clamps, if needed, to aid in Veress needle insertion, prior to initiating insufflation.
- TauTona Pneumoperitoneum Assist Device (TPAD): Participants receive investigational TPAD device during laparoscopic surgery prior to Veress needle entry and removed after insufflation is completed.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD)
Started | 15 | 16
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Count of Participants; unit: Participants]
  18-40 years old | 2 | 4 | 6
  41-64 years old | 9 | 3 | 12
  65 and over | 4 | 8 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 6 | 5 | 11
  White; Non-Hispanic/Non- Latino | 7 | 8 | 15
  Asian; Non-Hispanic/Non- Latino | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  18.5-24.9 kg/m^2 | 3 | 5 | 8
  25.0-29.9 kg/m^2 | 6 | 6 | 12
  30.0-34.9 kg/m^2 | 6 | 4 | 10
Skin Striae Severity [Count of Participants; unit: Participants] — Mild: Few striae, relatively small in size, and may be slightly discolored. Moderate: More numerous striae, slightly wider, and may be a more noticeable color.
  Severe: Many striae, wider, and may be a more prominent color (red, purple, or white).
  Extremely Severe: Extensive striae covering a large area, wide, and deeply colored (red, purple, or white).
  Participants
    None | 5 | 4 | 9
    Mild | 7 | 7 | 14
    Moderate | 2 | 3 | 5
    Severe | 1 | 1 | 2
    Extremely Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Satisfaction Survey
Description: The surgeon completes a LIKERT scale satisfaction survey related to the TPAD to assess its ease of use. Scale range 1-5 (higher scores correspond to higher satisfaction)
Time Frame: up to 1 minute on day of surgery
Population: Participants who completed the protocol
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD)
Number analyzed (Participants) | 15 | 15
score on a scale
  Obtaining counter traction for the Veress Needle was straightforward | 4 [3 to 4] | 4 [4 to 4]
  Advancing the Veress Needle into the peritoneal cavity was straightforward | 4 [3 to 4] | 4 [3 to 4]
  The Veress Needle was accurately inserted | 4 [3 to 4] | 4 [4 to 4]
  Advancing the Veress Needle into the peritoneal cavity was safe | 4 [3 to 4] | 4 [4 to 4]
  Inserting the Veress needle could be done by one physician | 4 [2 to 4] | 4 [3 to 4]
  Initiating and completing insufflation was straightforward | 4 [3 to 4] | 4 [3 to 4]

2. Secondary Outcome: Time From Incision for Veress Needle Insertion to Start of Insufflation
Time Frame: Up to approximately 2 minutes
Population: Participants who completed the protocol
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD)
Number analyzed (Participants) | 15 | 15
seconds | 87.0 [69.5 to 121.5] | 92.0 [81.5 to 127.5]

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: Adverse events related to use of the TPAD device
Time Frame: Continuous from start of surgery through postoperative day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD)
Number analyzed (Participants) | 15 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Standard of Care (SOC) | TauTona Pneumoperitoneum Assist Device (TPAD)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/16
Other Adverse Events (participants affected / at risk) | 14/15 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=15) | TauTona Pneumoperitoneum Assist Device (TPAD) (N=16)
Fluid Collection (Surgical and medical procedures) | 0 (0) | 1 (1) — Fluid collection in the gallbladder fossa with possible fistulization to the duodenum
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=15) | TauTona Pneumoperitoneum Assist Device (TPAD) (N=16)
Bruising (Surgical and medical procedures) | 14 (14) | 14 (14) — Bruising surrounding the Veress needle insertion site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04392635/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04392635/SAP_001.pdf